CLINICAL TRIAL: NCT01029158
Title: A Double-blind, Placebo Controlled, Randomised Trial to Compare the Efficacy of 250ng and 500ng RN1006 (a New Formulation of Avotermin) and 250ng and 500ng Juvista (Standard Avotermin Formulation), in the Improvement of Scar Appearance in Healthy Volunteer Subjects
Brief Title: A Trial to Compare the Efficacy of Two Formulations of Avotermin Against Placebo
Acronym: RN1006
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Renovo (Industry)
Responsible Party: Dr Jim Bush, Renovo
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: RN1006-0100
Record Dates: First submitted 2009-12-04; First posted 2009-12-09 (Estimated); Last update posted 2010-12-09 (Estimated); Status verified 2010-12

CONDITIONS: Scar Improvement
Keywords: Healthy volunteers; Comparison of two formulations; Improvement of scar appearance
MeSH Terms: interventions — TGFB3 protein, human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- 1a (Experimental): 250 ng Juvista or placebo injected intradermally down each 1 cm of wound margin immediately after wound closure. Then a further 250 ng Juvista or placebo injected intradermally down each 1 cm of wound margin 24 (+/- 4) hours after administration of the first dose.
  Interventions: Drug: Juvista (Avotermin); Drug: Placebo
- 1b (Experimental): 250 ng RN1006 or placebo injected intradermally down each 1 cm of wound margin immediately after wound closure. Then a further 250 ng RN1006 or placebo injected intradermally down each 1 cm of wound margin 24 (+/- 4) hours after administration of the first dose.
  Interventions: Drug: RN1006 (Avotermin); Drug: Placebo
- 1c (Experimental): 250 ng RN1006 or placebo injected intradermally down each 1 cm of wound margin immediately after wound closure.
  Interventions: Drug: RN1006 (Avotermin); Drug: Placebo
- 1d (Experimental): 500 ng RN1006 or placebo injected intradermally down each 1 cm of wound margin immediately after wound closure.
  Interventions: Drug: RN1006 (Avotermin); Drug: Placebo
- 2a (Experimental): 250 ng Juvista or placebo injected intradermally down each 1 cm of wound margin immediately after wound closure. Then 250 ng Juvista or placebo injected intradermally down each 1 cm of wound margin 24 (+/- 4) hours after administration of the first dose.
  Interventions: Drug: Juvista (Avotermin); Drug: Placebo
- 2b (Experimental): 500 ng Juvista or placebo injected intradermally down each 1 cm of wound margin immediately after wound closure.
  Interventions: Drug: Juvista (Avotermin); Drug: Placebo
- 2c (Experimental): 500 ng Juvista or placebo injected intradermally down each 1 cm of wound margin immediately after wound closure. Then a further 500 ng Juvista or placebo injected intradermally down each 1 cm of wound margin 24 (+/- 4) hours after administration of the first dose.
  Interventions: Drug: Juvista (Avotermin); Drug: Placebo
- 2d (Experimental): 500 ng RN1006 or placebo injected intradermally down each 1 cm of wound margin immediately after wound closure. Then 500 ng RN1006 or placebo injected intradermally down each 1 cm of wound margin 24 (+/- 4) hours after administration of the first dose (i.e. two doses in total).
  Interventions: Drug: RN1006 (Avotermin); Drug: Placebo

INTERVENTIONS:
Drug: Juvista (Avotermin) — 250 ng, twice, intradermal injection, standard formulation
  Other Names: juvista; RN1001
  Arms: 1a
Drug: RN1006 (Avotermin) — 250 ng, intradermal injection, twice
  Other Names: RN1006
  Arms: 1b
Drug: RN1006 (Avotermin) — 205 ng, Intradermal injection, once
  Other Names: RN1006
  Arms: 1c
Drug: RN1006 (Avotermin) — 500ng, intradermal injection, once
  Other Names: RN1006
  Arms: 1d
Drug: Juvista (Avotermin) — 250 ng, intradermal injection, twice
  Other Names: Juvista; RN1001
  Arms: 2a
Drug: Juvista (Avotermin) — 500 ng, intradermal injection, once
  Other Names: Juvista; RN1001
  Arms: 2b
Drug: Juvista (Avotermin) — 500 ng, intradermal injection, once
  Other Names: Juvista; RN1001
  Arms: 2c
Drug: RN1006 (Avotermin) — 500 ng, intradermal injection, twice
  Other Names: RN1006
  Arms: 2d
Drug: Placebo — Placebo

SUMMARY:
RN1006 has been developed as a stabilized formulation of avotermin which, when dosed once in pre-clinical studies in animals, has shown comparable scar improvement efficacy to the standard twice-dosed Juvista formulation. The aim of this trial is to investigate the efficacy of RN1006 compared to Juvista in a human volunteer model

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18-85 years who have given written informed consent
* Subjects with a body mass index within range 18-35 kg/m2
* Subjects with clinically acceptable results for the laboratory tests specified in the trial protocol
* Female subjects using a highly effective method (S) of contraception

Exclusion Criteria:

* Subjects who have a history of keloid scarring, surgery within one year of the first dosing area
* Subjects who have current scars, tattoos, birthmarks, mole within 3 cm of the area to be excised
* Subjects with any clinically significant medical condition or history of any condition which may impair wound healing

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2009-08; Primary Completion 2010-09 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Global scar comparison scale | 12 months

SECONDARY OUTCOMES:
Adverse event incidence including specific assessment of local tolerability at the treated wound site | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Renovo CTU, Manchester, United Kingdom